CLINICAL TRIAL: NCT04212624
Title: Clinical Research of Human Retinal Pigment Epithelial (HuRPE) Cell Injection on Atrophy of High Myopia Macular Area
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Eyecure Therapeutics Inc. (Industry)
Responsible Party: Principal Investigator, Xiaodong Sun, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JR-HuRPE-HMML-02
Record Dates: First submitted 2019-10-23; First posted 2019-12-27 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Degenerative Myopia With Macular Hole
Keywords: Human retinal pigment epithelial (HuRPE) cell injection; High myopia; retinal degeneration
MeSH Terms: conditions — Retinal Degeneration | interventions — Carboxylesterase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- test arm (Experimental): The 25G or 23G conjunctival seamless vitrectomy was performed on the anterior eye to remove the anterior-posterior direction and tangential direction of the rupture hole. The area outside the macular foveal lesion was selected, but 100 μl of HuRPE cell injection was injected within about 2 PD. In combination with the Medone syringe and the combined 35G or 37G needle, the silicone oil injection module is used for injection, and the injection is performed in an amount of 100 μl (depending on the cell concentration). The doses of the three dose groups from low to high were 300,000 cells, 500,000 cells, and 1 million cells, respectively, in a single injection.
  Interventions: Other: Human retinal pigment epithelial (HuRPE) cell injection

INTERVENTIONS:
Other: Human retinal pigment epithelial (HuRPE) cell injection — Human retinal pigment epithelial cell injection Dosage form and specifications: injection; 600,000 cells / branch (200μl), 1 million cells / branch (200μl), 2 million cells / branch (200μl) Transportation and storage: sealed, stored at 2-8 ° C, valid for 6 hours

SUMMARY:
To evaluate the safety and tolerability of human retinal pigment epithelial (HuRPE) cell injection subretinal transplantation for atrophy of high myopia macular area, and to explore the maximum tolerated dose (MTD).

DETAILED DESCRIPTION:
This study is a perspective, single-arm and open-labeled investigation of the safety and preliminary efficacy of unilateral subretinal transplantation of HuRPE cells in subjects with Macular degeneration caused by high myopia. The investigators will recruit and enroll 9 patients based on specific inclusive/exclusive criteria. Experimental and self-controlled eye will be determined based on best-corrected visual acuity (BCVA). The eye with BCVA between 5 and 60 ETDRS letters will be determined as experimental eye, which will be divided into 3 groups and undergo subretinal injection of 3 different dosages of HuRPE cells (300.000, 500,000 or 1,000,000) respectively, while the other one as control eye, will not receive the surgery.

HuRPE cells will be obtained from Eyecure Therapeutics, Inc.(Jiangsu) located in WuXi, Jiangsu Province. The obtained HuRPE cells will meet its quality standards and conform to Good manufacturing practices (GMP). HuRPE cells will be transplanted by a board-certified vitreoretinal surgeon, which will be administered into the subretinal space of experimental eye through a standard surgical approach.

Immunosuppressive agents will be administered orally to all subjects after transplantation. Dosage and time duration of immunosuppressive agents will be regulated strictly relying on the condition of immune rejection. Subjects will be monitored with ophthalmologic and systemic examinations frequently at regular post-transplant intervals after HuRPE cells transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. A patient who is able (or with the assistance of his or her legal representative) to read and understand the informed consent form and is willing to sign a written informed consent;
2. age ≥ 18 years old, male or female;
3. myopic diopter ≥ -6D or visual axis length ≥ 26mm;
4. study the best corrected visual acuity ≥ 5 letters, ≤ 60 letters (using ETDRS eye chart);
5. According to the researcher's judgment, the patient's high myopia macular atrophy is the main reason for the patient's vision loss;
6. If both eyes meet the inclusion criteria, the selected disease is more severe; the eyes are the same, and the right eye is the study eye.

Exclusion Criteria:

1. The study eye has intravitreal hemorrhage within 2 months before the group visit;
2. the study of the eye involved in the foveal scar, fibrosis, suggesting a serious irreversible vision loss;
3. The study eye diagnosis is a pupillary afferent defect (APD);
4. the study eye has significant refractive interstitial opacity, and moderate to severe cataract, may cause interference to OCT and fundus examination;
5. any eye diagnosed as infectious blepharitis, keratitis, scleritis or conjunctivitis; or there are currently serious systemic infectious diseases;
6. Uncontrollable glaucoma, defined as a patient who is adequately treated with medication, with an intraocular pressure still above 25 mmHg, or who has undergone previous or filtering surgery;
7. Study the eye with other diseases that affect vision;
8. traumatic macular hole, idiopathic macular hole, combined with other parts of the retinal tear;
9. single eye blind patients;
10. The study eye is an aphakic eye (except for the intraocular lens);
11. Any eye has a history of idiopathic or autoimmune-related uveitis;
12. Any eye is diagnosed as an iris neovascularization;
13. Received cataract surgery within 2 months prior to enrollment;
14. Other intraocular surgery was performed within 3 months prior to the group visit;
15. Have an allergic reaction or allergic history to sodium fluorescein, a history of allergies to protein products for therapeutic or diagnostic use, and allergies to two or more drugs and/or non-drug factors, or those with allergic diseases;
16. Diabetes patients with uncontrolled blood glucose (fasting blood glucose ≥7.0mmol/L or 2h postprandial blood glucose ≥11.1mmol/L);
17. There is a history of surgery within 1 month before screening, or there are currently unhealed wounds, ulcers, fractures, etc.;
18. patients with uncontrolled hypertension, defined as the best treatment plan, a single measurement of systolic blood pressure > 180mmHg, two consecutive measurements of systolic blood pressure > 160mmHg or diastolic blood pressure > 100mmHg;
19. History of myocardial infarction within 6 months prior to enrollment;
20. There is active diffuse intravascular coagulation or obvious bleeding tendency before screening. Anticoagulation or anti-platelet aggregation drugs are used in addition to aspirin/non-steroidal anti-inflammatory drugs within 14 days before screening;
21. Any clinical problem that cannot be controlled (such as severe mental, neurological, cardiovascular, respiratory, malignant, Parkinson's, Alzheimer's disease, etc.);
22. Women of childbearing age were positive in the screening visit pregnancy test. Women who wish to breastfeed during the study. All women of childbearing age (male and female) did not agree to take effective contraceptive measures (such as intrauterine devices, birth control pills or condoms) during the entire study period and within 30 days of the end of the visit period;
23. Patients who participated or are currently participating in other clinical studies within 30 days prior to screening;
24. Hemoglobin <100 g/L, blood Plt≤100×109/L, neutrophil count <1.0×109/L, ALT/AST> upper limit of normal value (ULN)×1.5, Cr>1.3 mg/dL;
25. Researchers believe that patients who are not eligible for inclusion, or other medical conditions, limit subject compliance, safety, or impact study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with Local and systemic adverse events | six months following transplantation
  Descriptive analysis of frequency and types of adverse events experienced by each subject during the study period.

SECONDARY OUTCOMES:
Mean change of Best-Corrected Visual Acuity (BCVA) | six months following transplantation
  Best-corrected visual acuity (BCVA) will be assessed in a sitting position using manifest refraction and ETDRS-like visual acuity testing charts. higher scores means improvement of patient's visual acuity.
Evidence of successful engraftment | six months following transplantation
  Structural evidence (OCT imaging, fluorescein angiography, slit-lamp examination with fundus photography) that HuRPE cells have been implanted in the correct location.
Change in NEI VFQ-25 Total Score | six months following transplantation
  National eye institute 25-item visual function questionnaire (NEI VFQ-25) is a condition-specific measure which was designed to capture the specific impact of vision loss on health-related quality of life (HRQoL). The calculation for NEI VFQ-25 sub-scale scores and total score was performed according to the "NEI VFQ-25 Scoring Algorithm - August 2000". The NEI VFQ-25 consists of a base set of 25 vision-targeted questions representing 11 vision-related constructs, plus an additional single-item general health rating question. All items are scored so that a high score represents better functioning. Each item is then converted to a 0 to 100 scale so that the lowest and highest possible scores are set at 0 and 100 points, respectively. In this format scores represent the achieved percentage of the total possible score, e.g. a score of 50 represents 50% of the highest possible score.

IPD SHARING:
Plan to Share IPD: No